CLINICAL TRIAL: NCT06660108
Title: BASES MOLECULAIRES DU DEVELOPPEMENT DU LANGAGE ORAL ET DES TROUBLES SPECIFIQUES ASSOCIES
Brief Title: MOLECULAR BASIS OF LANGUAGE DEVELOPMENT AND ASSOCIATED DISORDERS
Acronym: TSLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Imagine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C23-79; IDRCB (Other: 2024-A00519-38)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Developmental Language Disorder
MeSH Terms: conditions — Language Development Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DLD patient and relative (Other)
  Interventions: Genetic: blood draw

INTERVENTIONS:
Genetic: blood draw — Multiple blood draw for genomic and transcriptomic investigations

SUMMARY:
Developmental Language Disorder (DLD) refers to children who present with language difficulties that are not due to a known biomedical condition or associated with autism spectrum disorder (ASD) or intellectual disability. The prevalence of DLD is ~7%-8% or 2% if severe forms are considered.

However, the clinical heterogeneity of language disorders, the presence of co-morbidities and the inconsistent terminology used for many years have hindered research and clinical practice. Distinguishing sub-groups of children with language problems is crucial when tackling the underlying genetic causes of this disease. Recently, several studies using high-throughput sequencing have better define the genetic basis of CAS but such studies focusing on DLD are limited. The investigation of more homogeneous cohorts of individuals that clearly distinguish DLD cases, from ID and not including children with CAS should improve our understanding of the genetic basis of this disorder.

In this study, we aim to built and investigate a well-characterized cohort of DLD patients using pangenomic approaches to better define the molecular basis of this disorder. All individuals will be analyzed using chromosomal microarray analysis and whole genome sequencing. Multiple observations and preliminary results suggest strong links with the genetic basis of other neurodevelopmental disorders.

The goal is to identify CNV or SNV as causative allele or risk factor and already known to be involved in other neurodevelopmental disorders as well as potential new variants.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Eligible families included at least one child over five years old with a formal diagnosis of severe and isolated DLD according to Phase 2 CATALISE criteria . Patients have undergone age-appropriate speech, language and reading evaluations by a speech-language physician and cognitive evaluations by a neuropsychologist, as well as evaluation by a pediatric neurologist to identify co-occurring developmental disorders (ADHD, ASD…) and a medical geneticist for known genetic disorders and genetic testing recommendations. All children included received appropriate speech therapy for at least one year, with a progress report indicating the persistence of language difficulties.

Exclusion Criteria:

* Cognitive impairment with non-verbal intellectual quotient (IQ) below 2 SD assessed with the Wechsler Preschool and Primary Scale of Intelligence (WPPSI), or the Wechsler Intelligence Scale for Children (WISC-IV or V) according to the age-appropriateness, ASD, moderate to severe hearing loss, orofacial structural abnormalities, known neurological or genetic disorders at the initial assessment. None of the patients met the diagnostic criteria for CAS according to the ASHA (American Speech-Language-Hearing Association, 2007. Childhood apraxia of speech www.asha.org/policy).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Identification of CNV or SNV involved in neurodevelopmental disorders | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Sud Francilien, Corbeil-Essonnes
  - Raymond Poincaré- Garches, Garches
  - Hopital Necker, Paris

REFERENCES:
- [Derived] Ormieres C, Lesieur-Sebellin M, Siquier-Pernet K, Delplancq G, Rio M, Parisot M, Nitschke P, Rodriguez-Fontenla C, Bodineau A, Narcy L, Schlumberger E, Cantagrel V, Malan V. Deciphering the genetic basis of developmental language disorder in children without intellectual disability, autism or apraxia of speech. Mol Autism. 2025 Feb 13;16(1):10. doi: 10.1186/s13229-025-00642-8. PMID 39948625